CLINICAL TRIAL: NCT01299454
Title: A Single-dose, Open-label, Parallel Group, Matched Study Evaluating the Pharmacokinetics of Oral OPC-34712 Tablet in Subjects With Normal Hepatic Function and Hepatically Impaired Subjects
Brief Title: A Study Evaluating the of OPC-34712 in Subjects With Normal Hepatic Function and Hepatically Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 331-09-225
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

ARMS (4):
- Normal (Active Comparator)
  Interventions: Drug: OPC-34712
- Mild (Active Comparator)
  Interventions: Drug: OPC-34712
- Moderate (Active Comparator)
  Interventions: Drug: OPC-34712
- Severe (Active Comparator)
  Interventions: Drug: OPC-34712

INTERVENTIONS:
Drug: OPC-34712 — All groups will receive a single oral 2-mg OPC-34712 dose on Day 1 with 240 mL room temperature still water. Subjects will be administered the OPC-34712 dose in the fasted state (at least 8 hours of fasting) and no food will be allowed for 4 hours postdose. Water will be restricted as part of the dosing procedure from 1 hour prior to dosing and 2 hours post-dose.

SUMMARY:
The purpose of this study is to evaluate how much of the investigational product gets into the blood stream and how long the body takes to get rid of it when given to subjects with a range of liver impairment compared to subjects with normal liver function.

DETAILED DESCRIPTION:
This is a multi-center, open-label, parallel-arm study in 1 group of subjects with normal hepatic function and 3 groups of subjects with varying degrees of hepatic impairment (mild, moderate, and severe). Subjects will be confined to the clinic from Day -1 to Day 8. Subjects will be contacted via telephone 30 days (+ 2 days) after the last dose of study medication to assess any new or ongoing AEs and to record concomitant medications. All groups will receive a single oral 2-mg OPC-34712 dose on Day 1 with 240 mL room temperature still water. Subjects will be administered the OPC-34712 dose in the fasted state (at least 8 hours of fasting) and no food will be allowed for 4 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of non-childbearing potential ≥ 18 years of age
* Body weight within ± 30% of ideal body weight as defined in the 1983 Metropolitan Height and Weight Tables. Minimum body weight no less than 50 kg.
* Able to provide written, informed consent.
* Male and female subjects who are surgically sterile; female subjects who have been postmenopausal for at least 12 consecutive months; or male subjects who agree to remain abstinent or to practice double-barrier forms of birth control and refrain from sperm donation from Screening through 90 days from the last dose of study medication.

Inclusion Criteria for Hepatically Impaired Subjects Only:

* Hepatically impaired subjects with creatinine clearance (CLcr) > 30 mL/min.
* Subjects with hepatic impairment should have relatively stable hepatic function for the duration of the study, and otherwise be in generally good health.
* A clinical diagnosis of hepatic cirrhosis based on biopsy and/or clinical criteria.
* Child-Pugh Class A (mild), B (moderate), or C (severe)
* Hepatically impaired subjects may be taking medications, which in the opinion of the clinical investigator and sponsor, are believed to be therapeutic for the subjects.
* Hepatically impaired subjects may have a history of or current hepatitis or be carriers of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibodies (anti-HC).

Inclusion Criteria for Subjects with Normal Hepatic Function Only

* Must be in good health as determined by medical history, physical examination, ECG, serum/urine biochemistry, hematology, and serology tests.
* Normal renal function as evidenced by CLcr that is within 20% of normal for the age, sex, and weight of the individual.

Exclusion Criteria:

* History of drug and/or alcohol abuse within 2 years prior to Screening.
* History of acquired immunodeficiency syndrome or human immunodeficiency virus (HIV) antibodies.
* History of any significant drug allergy or known or suspected hypersensitivity.
* A positive urine alcohol test and/or urine drug screen for substance of abuse at Screening or upon admission to the study center.
* Subjects having taken an investigational drug within 30 days preceding study entry.
* Any history of significant bleeding or hemorrhagic tendencies. Subjects with a history of bleeding tendencies secondary to hepatic impairment will not be excluded.
* A history of difficulty in donating blood.
* The donation of blood or plasma within 30 days prior to dosing.
* Consumption of alcohol and/or food and beverages containing methylxanthines, grapefruit, grapefruit juice, Seville oranges, or Seville orange juice within 72 hours prior to dosing.
* Exposure to any substances known to stimulate hepatic microsomal enzymes within 30 days prior to Screening through the end of the study.
* Subjects who have supine, sitting, or standing blood pressure, after resting for ≥ 3 minutes, higher than 140/90 mmHg or lower than 100/50 mmHg.
* Subjects who have a supine pulse rate, after resting for ≥ 3 minutes, outside the range of 40 to 90 bpm.
* Previous exposure to OPC-34712.
* Subjects who are pregnant or breastfeeding.
* Subjects with a QTcF interval ≥ 450 msec.
* Subjects with PT greater than 2 times control. Subjects with hepatic impairment with prolonged PT will be excluded based on the PI's discretion.
* Subjects with hepatic carcinoma or porto-hepatic shunts that have been surgically created or planted.
* Partial thromboplastin time > 70 seconds.

Exclusion Criteria for Hepatically Impaired Subjects Only:

* History of serious mental disorder including subjects who are pre-encephalopathic or encephalopathic as assessed by the Child-Pugh score and/or the PI's judgment.
* Major surgery of the digestive tract.

Exclusion Criteria for Subjects with Normal Hepatic Function Only:

* Clinically significant abnormality in past medical history.
* History of or current hepatitis, or carriers of HBsAg and/or anti-HC.
* Use of prescription, over-the-counter, herbal medication or vitamin supplements within 14 days prior to dosing and antibiotics within 30 days prior to dosing.
* History of serious mental disorders.
* Major surgery of the digestive tract (excluding appendectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Study Site, Miami, Florida
  - Study Site, Minneapolis, Minnesota
  - Study Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 participants were screened; of these 45 participants were enrolled recruited at 3 study sites in the United States (US).
Groups:
- Mild Hepatic Impairment: Participants with mild hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 milligrams (mg).
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment (Child-Pugh classification scheme)received a single dose of oral brexpiprazole 2 mg.
- Severe Hepatic Impairment: Participants with severe hepatic impairment (based on Child-Pugh classification scheme) received a single dose of oral brexpiprazole 2 mg.
- Normal Hepatic Function: Participants with normal hepatic function (based on Child-Pugh classification scheme) received a single dose of oral brexpiprazole 2 mg.
Period: Overall Study
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Normal Hepatic Function
Started | 8 | 8 | 6 | 23
Completed | 8 | 8 | 6 | 23
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mild Hepatic Impairment: Participants with mild hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
- Severe Hepatic Impairment: Participants with severe hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
- Normal Hepatic Function: Participants with normal hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
- Total: Total of all reporting groups
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Normal Hepatic Function | Total
Number analyzed (Participants) | 8 | 8 | 6 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (7.3) | 57.8 (3.8) | 51.2 (4.4) | 56.2 (5.2) | 56.4 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 5 | 10
  Male | 5 | 6 | 6 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Unbound Brexpiprazole Area Under the Concentration Time Curve (AUC) Calculated to the Last Observable Concentration at Time t (AUCt,u)
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/Early termination (ET).
Time Frame: Day 1 to Day 8
Population: Pharmacokinetics (PK) set consisting of all evaluable brexpiprazole PK parameters from enrolled particpants who had evaluable plasma concentrations.
Measure: Mean (Standard Deviation); unit: nanograms.hours/mL (ng*h/mL)
Groups:
- Normal Hepatic Function Matched to Mild Hepatic Function; Normal Hepatic Function Matched to Severe Hepatic Function.: Participants with normal hepatic function received a single oral dose of brexpiprazole 2 mg.
  Each participant with normal hepatic function was matched to a participant with hepatic impairment by age (within the decile or ± 5 years, whichever was less), sex, and weight (± 15%). Participants with hepatic impairment and within 30% of their ideal body weight (minimum body weight of 50 kg) were enrolled.
- Normal Hepatic Function Matched to Moderate Hepatic Function.: Participants with normal hepatic function received a single oral dose of brexpiprazole 2 mg.
  Each participant with normal hepatic function was matched to a subject with hepatic impairment by age (within the decile or ± 5 years, whichever was less), sex, and weight (± 15%). Participants with hepatic impairment and within 30% of their ideal body weight (minimum body weight of 50 kg) were enrolled.
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
nanograms.hours/mL (ng*h/mL) | 5.95 (2.58) | 4.87 (1.78) | 5.41 (1.37) | 4.28 (1.95) | 3.27 (0.93) | 3.63 (1.54)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; The primary comparison was each hepatic disease group (mild, moderate or severe) versus the control (normal group). To compare the primary PK parameters between each hepatic disease group and the control group, the 90% confidence interval (CI) for the difference in the means of the log-transformed data was calculated using a mixed effect analysis of variance; Test type: Non-Inferiority or Equivalence — Bioequivalence was claimed for a PK parameter if the 90% CI for the ratio of the geometric means of a PK variable fell within the interval [0.5, 2.0]. Due to the nature of the normal-theory CIs, this approach was equivalent to carrying out two 1-sided tests of hypothesis at the 5% level of significance; Mixed effect analysis of variance; Geometric Mean Ratio = 1.166, 90% CI 2-sided [0.776 to 1.751] — Due to the nature of the normal-theory CIs, this approach is equivalent to carrying out two 1-sided tests of hypothesis at the 5% level of significance
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function Matched to Moderate Hepatic Function; The primary comparison was each hepatic disease group (mild, moderate or severe) versus the control (normal group). To compare the primary PK parameters between each hepatic disease group and the control group, the 90% CI for the difference in the means of the log-transformed data was calculated using a mixed effect analysis of variance; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 1.375, 90% CI 2-sided [0.915 to 2.066] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.929, 90% CI 2-sided [0.581 to 1.488] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Unbound Brexpiprazole AUC Calculated From Time Zero to Infinity (AUC∞,u)
Description: Blood samples were taken at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  AUC (0 - ∞)= AUC from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Day 1 to Day 8
Population: PK set consisting of all evaluable brexpiprazole PK parameters from enrolled particpants who had evaluable plasma concentrations.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Normal Hepatic Function Matched to Moderate Hepatic Function.; Normal Hepatic Function Matched to Severe Hepatic Function.: Participants with normal hepatic function received a single oral dose of brexpiprazole 2 mg.
  Each participant with normal hepatic function was matched to a participant with hepatic impairment by age (within the decile or ± 5 years, whichever was less), sex, and weight (± 15%). Participants with hepatic impairment and within 30% of their ideal body weight (minimum body weight of 50 kg) were enrolled.
- Severe Hepatic Function: Participants with severe hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment. | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 7 | 6 | 7 | 7 | 3 | 5
ng*h/mL | 8.59 (5.29) | 5.85 (3.11) | 8.50 (2.17) | 5.62 (3.13) | 3.49 (0.848) | 3.36 (0.871)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometic Mean Ratio = 1.255, 90% CI 2-sided [0.702 to 2.244] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment. vs Normal Hepatic Function Matched to Moderate Hepatic Function; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 1.727, 90% CI 2-sided [0.977 to 3.052] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Hepatic Function vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometic Mean Ratio = 1.041, 90% CI 2-sided [0.506 to 2.142] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Unbound Maximum Plasma Concentration of Brexpiprazole (Cmax,u)
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  Cmax,u is the highest measured unbound plasma concentration during the dosing interval.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Normal Hepatic Function Matched to Mild Hepatic Function.; Normal Hepatic Function Matched to Moderate Hepatic Function.; Normal Hepatic Function Matched to Severe Hepatic Function.: Participants with normal hepatic function received a single oral dose of brexpiprazole 2 mg.
  Each subject with normal hepatic function was matched to a subject with hepatic impairment by age (within the decile or ± 5 years, whichever was less), sex, and weight (± 15%). Subjects with hepatic impairment and within 30% of their ideal body weight (minimum body weight of 50 kg) were enrolled.
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
ng/mL | 0.104 (0.0259) | 0.114 (0.0270) | 0.0648 (0.0143) | 0.0779 (0.0224) | 0.0392 (0.0105) | 0.0760 (0.0258)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.904, 90% CI 2-sided [0.707 to 1.156] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function Matched to Moderate Hepatic Function; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.850, 90% CI 2-sided [0.665 to 1.087] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.531, 90% CI [0.399 to 0.705] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Area Under the Curve of Brexpiprazole Calculated to the Last Observable Concentration at Time t (AUCt)
Description: Blood samples were taken at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  AUCt= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t) The AUCt was estimated using the linear trapezoidal rule.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Severe Hepatic Impairment: Participants with normal hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
- Normal Hepatic Function Matched to Severe Hepatic Function.: Participants with normal hepatic function received a single oral dose of brexpiprazole 2 mg.
  Each participant with normal hepatic function was matched to a particpant with hepatic impairment by age (within the decile or ± 5 years, whichever was less), sex, and weight (± 15%). Participants with hepatic impairment and within 30% of their ideal body weight (minimum body weight of 50 kg) were enrolled.
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
ng*h/mL | 1271 (569) | 1145 (539) | 1213 (405) | 1048 (422) | 622 (163) | 817 (306)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; The secondary comparisons were each hepatic disease group (mild, moderate or severe) versus the control (normal group). To compare the secondary PK parameters between each hepatic disease group and the control group, the 90% CI for the difference in the means of the log-transformed data was calculated using a mixed effect analysis of variance; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 1.103, 90% CI 2-sided [0.774 to 1.573] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function Matched to Moderate Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 1.199, 90% CI 2-sided [0.841 to 1.710] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.790, 90% CI 2-sided [0.524 to 1.189] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Area Under the Concentration Time Curve of Brexpiprazole From Time Zero to Infinity (AUC∞)
Description: Blood samples were taken at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  AUC (0 - ∞)= AUC from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
  The AUC∞ was estimated using the linear trapezoidal rule
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Normal Hepatic Function Matched to Mild Hepatic Function.: Participants with normal hepatic function received a single oral dose of brexpiprazole 2 mg.
  Each participant with normal hepatic function was matched to a participant with hepatic impairment by age (within the decile or ± 5 years, whichever was less), sex, and weight (± 15%). Participant with hepatic impairment and within 30% of their ideal body weight (minimum body weight of 50 kg) were enrolled.
- Normal Hepatic Function Matched to Severe Hepatic Function.: Participants with normal hepatic function received a single oral dose of brexpiprazole 2 mg.
  Each participant with normal hepatic function was matched to a participant ith hepatic impairment by age (within the decile or ± 5 years, whichever was less), sex, and weight (± 15%). Participants with hepatic impairment and within 30% of their ideal body weight (minimum body weight of 50 kg) were enrolled.
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 7 | 6 | 7 | 7 | 3 | 5
ng*h/mL | 1827 (1103) | 1393 (881) | 1960 (579) | 1345 (697) | 831 (234) | 788 (230)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 1.241, 90% CI 2-sided [0.719 to 2.143] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function Matched to Moderate Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 1.604, 90% CI 2-sided [0.942 to 2.732] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 1.077, 90% CI 2-sided [0.540 to 2.146] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Maximum Plasma Concentration of Brexpiprazole (Cmax)
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  Cmax is the highest measured concentration of the drug during the dosing interval.
  Actual blood sample times were used for PK calculations. Values for Cmax and tmax were determined directly from the observed data.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
ng/mL | 22.9 (7.60) | 26.7 (9.09) | 14.6 (4.63) | 19.3 (4.98) | 7.65 (2.69) | 17.7 (7.38)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric mean ratio = 0.856, 90% CI 2-sided [0.691 to 1.059] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function Matched to Moderate Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.742, 90% CI 2-sided [0.599 to 0.918] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.451, 90% CI 2-sided [0.352 to 0.577] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time to Cmax of Brexiprazole (Tmax)
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  Tmax is the time taken to reach highest measured concentration of the drug during the dosing interval.
  Actual blood sample times were used for PK calculations. Values for Cmax and tmax were determined directly from the observed data.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
h | 3.50 [1.00 to 5.00] | 3.50 [2.00 to 5.00] | 4.50 [3.00 to 24.0] | 4.50 [1.00 to 6.00] | 5.00 [4.00 to 24.0] | 5.00 [2.00 to 6.00]

8. Secondary Outcome: Apparent Clearance of Brexpiprazole From Plasma After Extravascular Administration (CL/F)
Description: The value of CL/F (brexpiprazole only) was determined as Dose/AUC∞.
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h/kg
Groups:
- Normal Hepatic Function Matched to Mild Hepatic Function.: Participants with normal hepatic function received a single oral dose of brexpiprazole 2 mg.
  Each participant with normal hepatic function was matched to a participants with hepatic impairment by age (within the decile or ± 5 years, whichever was less), sex, and weight (± 15%). Partipants with hepatic impairment and within 30% of their ideal body weight (minimum body weight of 50 kg) were enrolled.
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 3 | 5
mL/h/kg | 24.5 (28.2) | 25.4 (12.3) | 13.8 (2.72) | 26.0 (19.2) | 28.2 (6.70) | 34.2 (16.3)

9. Secondary Outcome: Unbound Fraction of Brexpiprazole in Plasma (fu)
Description: Blood samples were taken at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % unbound drug in the urine
Groups:
- Mild Hepatic Function: Participants with mild hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
- Moderate Hepatic Function: Participants with moderate hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
Arm/Group | Mild Hepatic Function | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Function | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
% unbound drug in the urine | 0.472 (0.0840) | 0.451 (0.112) | 0.462 (0.0786) | 0.400 (0.0442) | 0.544 (0.186) | 0.450 (0.0795)

10. Secondary Outcome: Apparent Unbound Clearance of Brexpiprazole From Plasma After Extravascular Administration (CLu/F)
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  The value of CLu/F (brexpiprazole only) was determined as dose normalized unbound area under the concentration-time curve from time zero to infinity (Dose/AUC∞,u).
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Function | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 7 | 6 | 7 | 7 | 3 | 5
mL/h/kg | 5674 (7165) | 5730 (2944) | 3115 (494) | 6768 (5833) | 6598 (1182) | 7697 (2653)

11. Secondary Outcome: Terminal-phase Elimination Half-life of Brexpiprazole (t1/2,z)
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  The t1/2,z was determined as (ln2)/λz.
  Terminal-phase elimination half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Groups:
- Sever Hepatic Function: Participants with severe hepatic impairment (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
Arm/Group | Mild Hepatic Function | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Function | Normal Hepatic Function Matched to Moderate Hepatic Function. | Sever Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 7 | 6 | 7 | 7 | 3 | 5
h | 103 (51.1) | 64.7 (24.6) | 116 (25.8) | 64.2 (26.2) | 81.1 (17.1) | 51.4 (8.21)

12. Secondary Outcome: Renal Clearance (CLr) of Brexipiprazole
Description: Urine samples were taken at pre-dose and during the following increments: 0 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, and 144 to 168 hours postdose.
  The value of CLr was calculated as Ae,u/AUCt.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
mL/h/kg | 0.0468 (0.0353) | 0.0263 (0.0244) | 0.0360 (0.0286) | 0.0422 (0.0383) | 0.0402 (0.0872) | 0.0193 (0.0203)

13. Secondary Outcome: Cumulative Amount of Brexpiprazole Excreted Into the Urine (Ae,u)
Description: Urine samples were taken at pre-dose and during the following increments: 0 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, and 144 to 168 hours postdose.
  The value of Ae,u was calculated as the summation of urine concentration × urine volume from each collection interval
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Mild Hepatic Function | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Function | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
ng | 4511 (3808) | 1854 (1500) | 3522 (2740) | 3837 (3358) | 2090 (4699) | 1326 (1427)

14. Secondary Outcome: Fraction of Systemically Available Brexpiprazole Excreted Into the Urine (fe,u)
Description: Urine samples were taken at pre-dose and during the following increments: 0 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, and 144 to 168 hours postdose..
  The value of fe,u was calculated as 100 × Ae,u/Dose.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of drug in urine
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
% of drug in urine | 0.226 (0.190) | 0.0927 (0.0750) | 0.176 (0.137) | 0.192 (0.168) | 0.104 (0.235) | 0.0663 (0.0713)

15. Secondary Outcome: AUCt for DM-3411 Metabolite
Description: as for outcome 4
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
ng*h/mL | 380 (195) | 683 (246) | 284 (164) | 486 (263) | 151 (51.4) | 479 (226)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.509, 90% CI 2-sided [0.346 to 0.748]
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function Matched to Moderate Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.586, 90% CI 2-sided [0.399 to 0.861] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.334, 90% CI 2-sided [0.214 to 0.521] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: AUC∞ for DM-3411 Metabolite
Description: Blood samples were taken at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  The AUC∞ were estimated using the linear trapezoidal rule.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 4 | 3
ng*h/mL | 489 (210) | 692 (259) | 382 (262) | 530 (211) | 187 (67.2) | 329 (167)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.716, 90% CI 2-sided [0.445 to 1.153]
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function Matched to Moderate Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.594, 90% CI 2-sided [0.378 to 0.934]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.561, 90% CI 2-sided [0.308 to 1.022]

17. Secondary Outcome: Cmax for DM-3411 Metabolite
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET. Cmax is the highest measured concentration of the metabolite during the dosing interval.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
ng/mL | 6.49 (5.13) | 10.5 (4.26) | 3.19 (1.56) | 7.25 (4.83) | 2.15 (0.880) | 7.13 (3.73)
Statistical Analysis 1: Comparison: Mild Hepatic Impairment vs Normal Hepatic Function Matched to Mild Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.558, 90% CI 2-sided [0.368 to 0.845]
Statistical Analysis 2: Comparison: Moderate Hepatic Impairment vs Normal Hepatic Function Matched to Moderate Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.516, 90% CI 2-sided [0.341 to 0.781]
Statistical Analysis 3: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function Matched to Severe Hepatic Function; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed effect analysis of variance; Geometric Mean Ratio = 0.314, 90% CI 2-sided [0.195 to 0.507]

18. Secondary Outcome: Tmax for DM-3411 Metabolite
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET. Tmax is the time taken to reach highest measured concentration of the metabolite during the dosing interval.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Mild Hepatic Function | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Function | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
h | 5.00 [2.00 to 24.0] | 6.00 [5.00 to 24.0] | 5.00 [2.00 to 24.0] | 7.00 [2.00 to 24.0] | 4.5 [3.00 to 24.0] | 6.00 [5.00 to 16.0]

19. Secondary Outcome: t1/2,z for DM-3411 Metabolite
Description: Blood samples were taken at pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose/ET.
  The t1/2,z was determined as (ln2)/λz.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 4 | 3
h | 78.8 (37.6) | 59.7 (15.7) | 87.2 (45.7) | 62.0 (26.4) | 84.6 (12.0) | 56.1 (8.25)

20. Secondary Outcome: Ae,u for DM-3411 Metabolite
Description: as for outcome 13
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Mild Hepatic Function | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Function | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
ng | 67086 (25276) | 81148 (23188) | 68413 (16993) | 71353 (41630) | 48190 (14756) | 83604 (34907)

21. Secondary Outcome: fe,u for DM-3411 Metabolite
Description: Urine samples were taken at pre-dose and during the following increments: 0 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, and 144 to 168 hours postdose.
  The value of fe,u was calculated as 100 × Ae,u/Dose.
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % metabolite excreted in urine
Arm/Group | Mild Hepatic Function | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Function | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Function | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
% metabolite excreted in urine | 3.23 (1.22) | 3.91 (1.12) | 3.30 (0.819) | 3.44 (2.01) | 2.32 (0.712) | 4.03 (1.68)

22. Secondary Outcome: CLr for DM-3411 Metabolite
Description: as for outcome 12
Time Frame: Day 1 to Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Mild Hepatic Impairment | Normal Hepatic Function Matched to Mild Hepatic Function. | Moderate Hepatic Impairment | Normal Hepatic Function Matched to Moderate Hepatic Function. | Severe Hepatic Impairment | Normal Hepatic Function Matched to Severe Hepatic Function.
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 6 | 6
mL/h/kg | 2.67 (1.31) | 1.83 (0.828) | 3.96 (2.32) | 1.90 (0.568) | 4.08 (1.68) | 2.33 (1.01)

23. Secondary Outcome: Number of Adverse Events (AEs) Reported
Description: AEs were captured for all participants from the time the ICF was signed until the end of the study
Time Frame: From the time the Informed Consent Form was signed, throughout the 8 day study up to 30 days after study drug administration.
Population: Participants who received at least one dose of study drug were included in the safety analysis.
Measure: Number; unit: Events
Groups:
- Normal Hepatic Function: Participants with normal hepatic function (Child-Pugh classification scheme) received a single oral dose of brexpiprazole 2 mg.
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 6 | 23
Events
  Adverse events | 3 | 5 | 1 | 8
  Treatment emergent adverse events | 3 | 5 | 1 | 6
  Serious adverse events | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With Changes From Baseline in Vital Signs Parameters.
Description: Vital signs (including blood pressure, heart rate, temperature, and respiratory rate) were assessed at Screening, Day -1, Day 1 at predose (within 45 minutes prior to dosing), and 2, 4, 6, 8, 12, 24, 72, 120, and 168/ET hours postdose. Blood pressure and heart rate were taken with the subject in the supine (performed first), sitting, and standing
Time Frame: Day -1 to Day 8
Population: The abnormal values of vital signs values in participants are captured as serious AEs/AEs and are reported in the SAE or other AE section of this results report.
Measure: Number; unit: Participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 6 | 23
Participants | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Changes From Baseline in Electrocardiogram (ECG) Parameters.
Description: Electrocardiograms were performed at Screening, Day -1, and Day 1 at predose (in triplicate; within 45 minutes prior to dosing), and 2, 4, 6, 8, 12, 24, 72, 120, and 168/ET hours postdose. Standard 12-lead ECGs were performed after the subject was supine and at rest for ≥ 10 minutes prior to the ECG.
Time Frame: Day-1 to Day 8
Population: The abnormal values of ECG values in participants are captured as serious AEs/AEs and are reported in the SAE or other AE section of this results report.
Measure: Number; unit: Participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 6 | 23
Participants | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Changes From Baseline in Serum Chemistry, Hematology and Urinalysis Parameters.
Description: Hematology, serum chemistry, and urinalysis, including prothrombin time, international normalized ratio, partial thromboplastin time, and activated partial thromboplastin time, were completed at Screening, Day -1, Day 3 (48 hours postdose), and Day 8 (168 hours postdose)/ET.
Time Frame: Day -1 to Day 8
Population: The abnormal values of laboratory values in participants are captured as serious AEs/AEs and are reported in the SAE or other AE section of this results report.
Measure: Number; unit: Participant
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 6 | 23
Participant | 0 | 0 | 0 | 0

27. Secondary Outcome: Incidence of Suicidality, Suicidal Behaviour or Suicidal Ideation as Measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Baseline version of the C-SSRS was administered at Screening. The Since Last Visit version of the C-SSRS was administered on Day 1 at predose and on Days 4 and 7.
Time Frame: Day 1, Day 4, Day 7
Population: Suicidality, suicidal behaviour or suicidal ideation are captured as serious AEs/AEs and are reported in the SAE or other AE section of this results report.
Measure: Number; unit: Participants
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 6 | 23
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time the Informed Consent Form was signed, throughout the 8 day study up to 30 days after study drug administration.
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Normal Hepatic Function
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/6 | 0/23
Other Adverse Events (participants affected / at risk) | 3/8 | 3/8 | 1/6 | 6/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mild Hepatic Impairment (N=8) | Moderate Hepatic Impairment (N=8) | Severe Hepatic Impairment (N=6) | Normal Hepatic Function (N=23)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 4
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No